CLINICAL TRIAL: NCT01004666
Title: Molecular Breast Imaging: A Novel Technology for Detection of Malignant Breast Lesions.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-09-EE-0192-CTIL
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Small Breast Lesions; Dense Breast Tissue; Discrepancy With Clinical Examination; Equivocal Mammographic, Sonographic or MRI Lesion
Keywords: Breast cancer; Scintimammography; CZT; High-risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Women with equivocal findings on Mammography, US and/or MRI: Women with equivocal findings on Mammography, US and/or MRI
- Discrepancy between clinical examination and imaging: Women with discrepancy between clinical examination and breast imaging
- Women with dense breast: Women with dense breast
- Women in high risk for Breast Cancer: Women in high risk for Breast Cancer. Including patients with genetic high risk and/or strong family history.

SUMMARY:
Detection of breast cancer as early as possible is an ongoing imaging challenge.The purpose of the current study is to assess the clinical performance of the new scintigraphic technology, a dedicated breast gamma camera composed by the new generation of CZT detectors,for assessment of breast pathology specifically in women where current imaging techniques, mainly mammography are suboptimal. These cohort are patients with dense breast tissue and patients who are at high risk for breast cancer by a combination of other metrics, including family history and genetic testing. BRCA (breast cancer susceptibility gene), is particularly a relevant health problem among Ashkenazi Jews in Israel.

DETAILED DESCRIPTION:
Recently, a breast-dedicated gamma camera has been used for assessment of breast malignancy in over 1000 women in Mayo Clinic, Rochester, USA. Molecular Breast Imaging (MBI), which utilizes a Cadmium-Zinc-Telluride (CZT) gamma camera for scintimammography, has been shown to have a high sensitivity (91%) for the detection of breast lesions > 5 mm in diameter and 69% for tumors smaller than 5mm.

In Israel , genetic high- risk for breast cancer is highly relevant. We will offer the new imaging technology, to a wide patients population/group from all over Israel , in which the referring physician and/or the breast-imaging physician will look for additional imaging modality. Therefore this stage will include:

* Women with equivocal findings on Mammography, US and/or MRI
* Women with discrepancy between CBE(clinical breast examination)and breast imaging
* Women with dense breast
* Women in high risk for Breast Cancer

Before the imaging procedure each woman will need to fill detailed questionnaire, specific for the study, that will include information on her medical history, family history, gynecology information, menstrual phase, use of hormones etc.

The images will be correlated with other imaging tests including mammography, US and MRI. We will follow up the women for at least 6 months, including biopsy findings and or other clinical and imaging exams.

This phase will include 500 women.

ELIGIBILITY:
Inclusion Criteria:

* Age over 25.
* Equivocal breast lesions.
* Dense breast tissue.
* High-risk for breast cancer

Exclusion Criteria:

* Age under 25.
* Pregnancy.
* Patients unable to understand and sign an informed consent

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A wide COHORT from all over Israel , in which the referring physician and/or the breast-imaging physician will look for additional imaging modality. Women with equivocal findings on Mammography, US and/or MRI. Women with discrepancy between clinical examination and conventional breast imaging. Women with dense breast. Women with genetic and/or family history high risk for Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Detection of unexpected malignant lesions. Ruling out malignant lesions in case of equivocal lesions identified by clinical examination, mammography, US and/or MRI. | 6 mounth post scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Einat Even-Sapir, MD, PhD, Principal Investigator — Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
Locations (1):
- Department of Nuclear Medicine, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Hruska CB, Phillips SW, Whaley DH, Rhodes DJ, O'Connor MK. Molecular breast imaging: use of a dual-head dedicated gamma camera to detect small breast tumors. AJR Am J Roentgenol. 2008 Dec;191(6):1805-15. doi: 10.2214/AJR.07.3693. PMID 19020253
- [Background] Hruska CB, Boughey JC, Phillips SW, Rhodes DJ, Wahner-Roedler DL, Whaley DH, Degnim AC, O'Connor MK. Scientific Impact Recognition Award: Molecular breast imaging: a review of the Mayo Clinic experience. Am J Surg. 2008 Oct;196(4):470-6. doi: 10.1016/j.amjsurg.2008.06.005. Epub 2008 Aug 23. PMID 18723155
- [Background] Hruska CB, O'Connor MK. Quantification of lesion size, depth, and uptake using a dual-head molecular breast imaging system. Med Phys. 2008 Apr;35(4):1365-76. doi: 10.1118/1.2885371. PMID 18491531